## Increasing Physical Activity Among Sedentary Older Adults: What, Where, When, and With Whom

NCT03124537

**Informed Consent** 

Upload Date: 05/13/2020 Document Date: 10/3/2018







## **Informed Consent StepMate Walking App Study**

This research study, which is conducted by the Boston Roybal Center for Active Lifestyle Interventions at Brandeis University, is about using a new app, StepMate to help you increase your physical activity by walking. There are three components to this study: answering questionnaires through the internet, mail, and/or phone, using the new app on your iPhone on a daily basis, and increasing the number of daily steps over a one month period. Upon completing the study, you will receive a \$25 Amazon.com e-gift card. In addition, you will be able to keep the app in appreciation for your participation.

This study will take place over the course of one month. The study can be done at home; you do not need to come to the university. At the beginning and end we will ask you to fill out a series of questionnaires. Completing the questionnaires at each of the two occasions (at the beginning and end of the study) should take about 30 minutes each time, and you can do this in your own home at times that are convenient for you. You will also be given the app to download on your smartphone, which you may keep upon completion of the study. We would like you to check the app each day and to respond to the brief questions that you will receive a few times each day from the app. At the end of the one-month period, you will be asked again to fill out the questionnaires, at a convenient time.

The walking app has multiple components, all of which are aimed at helping you to increase the number of steps you walk each day. Persons enrolled in the study will get different versions of the app. The goal for us is to compare the different versions of the app to see which aspects are the most helpful for increasing activity levels. Any risks involved in this study are minimal and no greater than those encountered in everyday life. It is possible, although unlikely, that some participants may experience an injury or become physically fatigued from engaging in an increased amount of activity.

The direct personal benefits associated with participating in this study include receiving the app to keep upon completion of the study. You will also receive a \$25 Amazon.com e-gift card.

If you increase your physical activity you may also experience benefits to your overall health. The information collected by the researchers will be entirely confidential and will be used for research purposes only. Your name will not be used in any reports and all of your responses, including the information provided by internet, phone calls, and the app will be identified by a number and not your name. Data for all participants will be combined and analyzed as a group. Therefore, we will not be able to give you specific feedback about your individual results. Upon request, we will be happy to send you a summary of the overall research findings when they are available.

To help protect your privacy, this research is covered by a Certificate of Confidentiality. This means that the researchers may not disclose or use any information that may identify you unless you have consented to its use. Information or documents protected by this Certificate cannot be disclosed to anyone who is not connected with the research, unless there is a law that requires disclosure; if you have consented to the disclosure; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects. A Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want

## **Brandeis University**



Lifespan Developmental Psychology Lab Mailstop 062 participate.stepmate@gmail.com 781-736-3284



your research information released to any person not connected with the research, you must provide specific information about what you want the researchers to release.

Your participation in this study is voluntary; and you are completely free to withdraw from the study at any time or to refuse to answer any questions, or to decline participation in any component of the study. If you do not complete the study, you will still be able to keep the app.

By signing below, you state that you have heard and understand the explanation of this study and freely consent to participate in it; that you understand that your participation is voluntary; and that you are completely free to withdraw from the study at any time or to refuse to answer any questions, or to decline participation in any component in the study.

By signing below, you agree that all questions you may have had about the study have been explained to your full satisfaction. If you have further questions about the study, you may contact the Principal Investigator, Margie Lachman, or her research assistant at the Lifespan Lab 781 736 3284. If you have questions about your rights as a research subject please contact the Brandeis Institutional Review Board at irb@brandeis.edu or 781-736-8133.

| Participant's name (please print): | |
|---|---|
| Participant's signature: | Date: |
| Researcher's signature: | Date: |
| Please sign and return this form using the enclosed stamped an Boston Roybal Center for Active Lifestyle Interventions Lifespa Brandeis University Brown Social Sciences Building Psychology Department MS 062415 South Street | n Lab |
| Waltham, MA 02454 | |